CLINICAL TRIAL: NCT00003664
Title: Combination Chemobiotherapy With Gemcitabine, 5-Fluorouracil, Interleukin-2 and Alpha Interferon in Patients With Metastatic or Unresectable Renal Cell Cancer. A Phase II Study
Brief Title: Combination Chemotherapy and Biological Therapy In Treating Patients With Kidney Cancer That Is Metastatic or Cannot Be Removed Surgically
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Biotherapy Research Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066757; CBRG-9808; NCI-V98-1493
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2000-09

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha; Fluorouracil; Gemcitabine

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Drug: fluorouracil
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill kidney cancer cells. Interferon alfa may interfere with the growth of cancer cells. Combining chemotherapy with biological therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and biological therapy in treating patients with kidney cancer that is metastatic or cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effects of interferon alfa, interleukin-2, gemcitabine, and fluorouracil in patients with metastatic or unresectable renal cell cancer. II. Evaluate the feasibility and possible therapeutic anticancer efficacy of this therapy in these patients. III. Determine the duration of response, survival, and improvement of quality of life in these patients.

OUTLINE: Patients receive fluorouracil IV on days 1, 8, 15, and 22, followed by gemcitabine IV over 30 minutes on days 29, 36, 43, and 50. Interferon alfa is administered subcutaneously 3 times weekly beginning on day 1. Beginning on day 2, interleukin-2 is administered subcutaneously 3 times weekly for the first 4 weeks of the treatment course. Treatment is repeated every 8 weeks for up to 4 courses in the absence of unacceptable toxic effects and disease progression. Following chemobiotherapy, maintenance therapy is administered to patients with stable or responding disease. Patients receive subcutaneous interferon alfa 3 times weekly at the maximum tolerated dose until disease progression or for a maximum of 1 year. A quality of life assessment is completed weekly. Patients are followed until death.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic or unresectable carcinoma of the kidney No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: ECOG 0-2 Life expectancy: Greater than 4 months Hematopoietic: WBC at least 3,500/mm3 Granulocyte count at least 2,500/mm3 Platelet count at least 100,000/mm3 PT no greater than 1.3 times upper limit of normal (ULN) Hematocrit at least 28% Hepatic: Bilirubin less than 2.0 mg/dL SGOT no greater than 1.25 times ULN (unless due to tumor) Renal: Creatinine less than 2.0 mg/dL Calcium less than 12 mg/dL Proteinuria no greater than 2.0 by dipstick Cardiovascular: No active angina No uncontrolled congestive heart failure No uncontrolled arrhythmias No myocardial infarction within 6 months Pulmonary: No significant pulmonary disease (RA pO2 less than 60 or pCO2 greater than 50) Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative No active infection No daily emesis or inability to tolerate solid foods No prior or concurrent second malignancy within 2 years, except: Nonmelanoma skin cancer Carcinoma in situ of the cervix No sever diarrhea (greater than 4 watery stools per day) No active pelvic inflammatory disease No inflammatory bowel disease No uncontrolled seizure disorders No personal or family history of malignant hyperthermia No recent thromboembolism or any condition requiring concurrent anticoagulation

PRIOR CONCURRENT THERAPY: Biologic therapy: No other concurrent biologic therapy Chemotherapy: No prior gemcitabine No prior fluorouracil other than adjuvant fluorouracil received at least 1 year prior to study No other concurrent chemotherapy Endocrine therapy: Concurrent corticosteroids not allowed (except for nausea or vomiting) Radiotherapy: At least 14 days since prior radiation to axial skeleton No concurrent radiotherapy (except to local lesions) Surgery: At least 14 days since prior exploration and biopsy At least 21 days since prior resection with anastomosis No major organ allograft Other: No concurrent barbiturates No concurrent oral anticoagulants No other concurrent investigational drugs or devices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-10

CONTACTS AND LOCATIONS:
Overall Officials: Gamini S. Soori, MD, FACP, FRCP, MBA, Study Chair — Cancer Biotherapy Research Group
Locations (2):
- United States (2):
  - Bloomington Hospital, Bloomington, Indiana
  - Bergan Mercy Medical Center, Omaha, Nebraska